

Subject Consent Form for Participation in Human Research at Montana State University

# Would you like to participate in the Messengers for Health Báa nnilah project?

# Why are you being asked to participate in the Báa nnilah project?

- This is a research project to teach Crow men and women about ongoing health concerns. The project will give you the opportunity to discuss your experiences and knowledge about ongoing health concerns.
- The goal of the project is to increase the amount of information that Crow men and women have about ongoing health concerns and to increase the number of men and women who take steps to keep themselves healthy. This could mean improving the health and wellness of Crow families. Community members who have an ongoing illness and who are 25 years old and older are welcome to participate.

### What will you be asked to do? How much time will it take?

- Participation is voluntary. If you choose to participate in the project, you will:
  - o Come to an orientation meeting for the program. The meeting will last 2-3 hours, held in a community on the reservation (Wyola, Pryor, Lodge Grass, Crow Agency) or in Hardin and be led by project staff members including Alma McCormick and Lucille Other Medicine. During the meeting, we will have a meal, share information about the program, take a survey that asks questions about ongoing health concerns, and perform 3 exercises including walking for 6 minutes, standing up from a chair and walking 10 feet and walking back to the chair to sit, and standing for balance. These exercises will be used to develop an exercise program for you. For the survey, a member of the Báa nnilah team will read the survey questions to you and you will enter your answers on a computer privately so that no one will see your answers. You will come to another group meeting where you will take the same survey and complete the same exercises 4 times over the next 18 months.
  - o Fill out a form that lists your ongoing health concerns.
- o Attend 7 gatherings with about 10 other people where you will learn about ongoing health concerns. These gatherings will take place in local communities (Wyola, Pryor, Lodge Grass, Crow Agency, Hardin) and be led by a community mentor. Each of the 7 gatherings will last for 3 hours and include a meal and hands-on activities. Project staff members such as Alma McCormick and Lucille Other Medicine may late approved also attend the gatherings.



o 20 participants will also be asked to complete an hour-long interview with Alma McCormick or another staff member after the gatherings are completed. The interview will help us to make the Báa nnilah program better for the future.

# Do you have to take the survey or do the exercises?

No. You do not have to take the survey or do the exercises. Participation is voluntary and you can choose to not answer any questions you do not want to answer and/or you can stop anytime. There will be no penalty if you decide not to take the survey or do the exercises.

#### How did you get my name for this survey?

You expressed interest in participating in the Báa nnilah project. You may have met with a project mentor or staff member in the community.

### Are there any risks involved with taking part in the project? Will you feel uncomfortable?

- Taking part in the project should not put you at risk for physical harm. You may feel uncomfortable answering certain questions on the survey. You can perform the 3 exercises as you feel comfortable. You will never be required to answer any questions that make you feel uncomfortable or do any exercises that you do not want to do.
- During one of the gatherings, there will be a discussion of grief, loss, resilience, and healing. You will be provided with a list of resources available in the local communities for you to access if you desire.
- In the event your participation in this research supported by the National Institutes of Health results in injury to you, medical treatment consisting of a referral to Indian Health Services or Bighorn Valley Health Center will be available. If it is an emergency, a project mentor or staff member will call 911. This treatment will be at your expense. Further information about this treatment may be obtained by calling Alma McCormick at 665-5492 or Suzanne Held at Montana State University at 994-6321.

# What will you get out of taking part in the project? Will you get paid?

- You will be provided with a \$40.00 gift card each time you come to the meeting where you will complete the survey and exercises. This is to thank you for taking your time to do these things. You will also help us learn about ongoing health concerns among women and men in the Crow community. This information will help us learn if our Báa nnilah program is helping people and how to make it better for others.
- At each of the 7 gatherings, you will also receive a meal, incentives that encourage healthy living, and a \$10 gas card to help with transportation to the gatherings.

Is there any cost for you to participate in the Báa nnilah program?

No, there is no cost for you to participate in the program.



#### Will people know that you took part in the project?

- To ensure confidentiality, you will be entering your answers to the survey into a computer tablet. The tablet does not have your name included. The information from the computer tablets will be transferred securely and stored on computers that have a password that only people working on this project can have access to. The mentors and project staff who will be giving you the survey have signed a form agreeing not to share any information.
- This project is a clinical trial. A description of the clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search the Web site at any time.

#### Who is paying for this project?

The National Institutes of Health is paying for this project.

## Why do you have me signing this form?

This type of form is used any time people gather information for a research project. It is done to make sure that you understand any risks of taking the survey and completing the exercises and to give you people to contact in case you have any questions about the Báa nnilah project.

# What if you have any questions about the project or your participation?

If you ever have any questions about this project, please feel free to contact the project coordinator, Alma McCormick at 665-5492 or Suzanne Held at Montana State University at 994-6321.

# What if you have any questions about your rights regarding this project?

If you ever have any questions about your rights, you can contact Mark Quinn, the Chair of the Human Subjects Committee at Montana State University. His number is (406) 994-5721.



If you are interested in being a part of the Báa nnilah project, please read the following agreement statement and sign your name below the statement.

# Agreement statement:

| , , , | o participate in the Báa nnilah project. I |
|---|---|
| | nderstand the discomforts, inconvenience, (name of participant) agree to |
| be a part of the Báa nnilah project. I uparticipate, and that I may withdraw freceived a copy of this consent form f | rom the project at any time. I have |
| Participant signature | Date |
| Mentor Signature | Date |

